CLINICAL TRIAL: NCT04493125
Title: The Effect of Mosapride Citrate on Gastrointestinal Motility After Laparoscopic Gastrectomy: Prospective, Double Blind Placebo-controlled Study
Brief Title: Effect of Mosapride Citrate on Gastrointestinal Motility After Laparoscopic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Assistnat Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2020-0175
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Stomach Cancer
Keywords: Gastrectomy, Intestinal motility, Mosapride, Adhesion, Ileus
MeSH Terms: conditions — Stomach Neoplasms; Tissue Adhesions; Ileus | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mosapride group (Experimental): Patients receive placebo or mosapride citrate (5mg/T) three times a day from the first day after surgery.
  Interventions: Drug: Mosapride citrate
- Placebo group (Placebo Comparator): Patients receive placebo instead of mosapride citrate (5mg/T) three times a day from the first day after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mosapride citrate — Patients receive mosapride citrate (5mg/T) three times a day from the first day after surgery.
  Arms: Mosapride group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
"Mosapride citrate is a 5-hydroxytryptamine 4 receptor agonist, and is widely used as an agent to increase intestinal motility. Mosapride citrate has been demonstrated in in vitro and in vivo studies to increase both gastric and colon motility. In a case-control study of patients undergoing colonectomy, mosapride citrate was found to significantly reduce gas passing and defecation time.

Recently, a study reported that mosapride citrate acts on the α7nACh receptor and, consequently, suppresses the inflammatory response of macrophages, thereby suppressing the mechanism that induces paralysis after surgery.

To date, this study is intended to analyze whether mosapride citrate significantly affects the improvement of bowel movement after surgery after gastrectomy."

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with gastric cancer pathologically before surgery
2. Patients who underwent surgical resection (R0 resection)
3. Patients with an ASA score of 3 or less

Exclusion Criteria:

1. Patients over 80 years old
2. When there are multiple or peritoneal metastases
3. Intestinal obstruction before surgery
4. When chemotherapy was performed before surgery
5. When cancer other than stomach cancer is diagnosed
6. If you have a long history of major intra-abdominal surgery or a history of abdominal radiotherapy
7. In case of liver failure or kidney failure
8. When it is judged that uncontrolled diabetes may affect intestinal function

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
The number of radiopaque markers transferred to the large intestine 3 days after surgery | 3 Days after surgery
  Intestinal motility after gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea